CLINICAL TRIAL: NCT02259075
Title: Botulinum Toxin Type A Block of the Sphenopalatine Ganglion in Chronic Migraine. Safety Issues.
Brief Title: Botox Injection in Treatment of Chronic Migraine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTACM2014; 2014-001852-43 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Migraine Disorders
Keywords: Migraine with aura; Migraine without aura; Headache disorders; Botulinum Toxin Type A; Sphenopalatine Ganglion Block; Autonomic Nerve Block
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botulinum Toxin (Experimental): The patients will be injected with 25 IU of Botulinum Toxin Type A towards both the right and left sphenopalatine ganglion, a total of 50 IU.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Other Names: Botox; BTA

SUMMARY:
Chronic migraine is in many cases a most disabling condition. Chronic migraine is defined as headaches for at least 15 days per month, of which 8 days have typical migraine features. In many cases, oral drug treatment has little effect.

The parasympathetic nervous system acting through the sphenopalatine ganglion may be involved in several primary headaches, including migraine, by facilitating release of inflammatory substances in cerebral vessels. Botulinum toxin type A (BTA) inhibits excretion of acetylcholine resulting in blocking of nerve signals in the sphenopalatine ganglion.

The purpose of the present study is to evaluate a new technique with injection of BTA using an minimal invasive image guided procedure, for blocking of the sphenopalatine ganglion. The goal is to relieve the migraine symptoms and develop an alternate treatment for cases where oral drug treatments fail.

The main objective of the project is to determine the safety of this method of BTA injection in the area of the sphenopalatine ganglion by detecting adverse events. Secondary objectives are to measure changes in headache attack parameters with this novel method.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Chronic migraine with or without aura defined in International Classification of Headache Disorders (ICHD)-3 criteria
* Failed at least 3 oral migraine prophylactic treatments
* Duration of migraine at least 1 year before inclusion
* Start of migraine before participant turned 50 years
* Participant can make a distinction between migraine and other types of headache

Exclusion Criteria:

* If the criteria for medication-overuse headache (MOH) is fulfilled
* Heart or lung disease
* Any kind of systematic or local disease or illness that may significantly increase the risk of complications for the procedure related to injection
* Psychiatric illness that hinders participation in the study
* Known pregnancy or breast feeding
* Inadequate use of contraceptives
* Overuse or abuse of opioids
* Abuse of medications, narcotics or alcohol
* Anomalies which hinder or impede the used method of injection
* Allergy or any other hypersensitivity reactions against marcain, lidocaine, xylocain or adrenalin, botulinum toxin type A, Botox or any of it's constituents or any other related medication
* Treatment with medication that can interact with botulinum toxin type A

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and number of participants with adverse events | For the follow-up period of 3 months
  Number of adverse events and number of participants with adverse events after BTA injection in the area of the sphenopalatine ganglion and severity of adverse events by the method used. Registration of any adverse events categorized by probable relationship to drug or the procedure. Data obtained from the headache diaries as well as open questions during consultations.
Number of headache days with moderate or severe intensity | 5-8 weeks
  measured from week 5 to week 8, in total during 4 weeks

SECONDARY OUTCOMES:
Number of reponders | 12 weeks
  response is defined as ≥ 50% reduction in number of headache days with moderate or severe intensity per 4 weeks (week 1-4, week 5-8, week 9-12)
Days with moderate or severe headache per 4 weeks | 12 weeks
  week 1-4, week 5-8, week 9-12
Days without headache per 4 weeks | 12 weeks
  week 1-4, week 5-8, week 9-12
Hours with headache of moderate or severe headache per 4 weeks | 12 weeks
  week 1-4, week 5-8, week 9-12

CONTACTS AND LOCATIONS:
Overall Officials: Erling A Tronvik, PhD, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Bratbak DF, Nordgard S, Stovner LJ, Linde M, Dodick DW, Aschehoug I, Folvik M, Tronvik E. Pilot study of sphenopalatine injection of onabotulinumtoxinA for the treatment of intractable chronic migraine. Cephalalgia. 2017 Apr;37(4):356-364. doi: 10.1177/0333102416648328. Epub 2016 May 6. PMID 27154997